CLINICAL TRIAL: NCT04595513
Title: Stopping TSC Onset and Progression 2: Epilepsy Prevention in TSC Infants
Acronym: STOP2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-1045
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Tuberous Sclerosis Complex; Epilepsy
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: This trial is a single stage, phase I/II clinical trial design. Treatment is open-label to verify safety and dosing for TAVT-18 in TSC infants.
  Note that this clinical trial originally planned for a follow-up second stage employing a randomized, double-blind, placebo-controlled multisite design. In October 2021, the second stage of this study was replaced by the TSC-STEPS clinical trial (clinicaltrials.gov NCT05104983).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stage 1 Open Label (Experimental): Phase I/II, open-label PK and initial safety analysis. TAVT-18 administered orally twice/daily to achieve precision dosing target of 10 ng/ml. Whole blood sirolimus levels are assessed at defined intervals on days 1, 7, and 14. After day 14, participants can elect to continue open-label treatment with TAVT-18 until 12 months of age. Final developmental outcomes are assessed at 24 months of age.
  Interventions: Drug: TAVT-18 (sirolimus)

INTERVENTIONS:
Drug: TAVT-18 (sirolimus) — The investigational drug product to be used in this study is TAVT-18, a proprietary formulation of sirolimus in clinical development, by Tavanta Therapeutics, Inc. It is provided in a powder formulation in pre-measured vials.

SUMMARY:
This phase I/II clinical trial is an open-label clinical trial design to verify safety and dosing for TAVT-18 (sirolimus) powder for oral solution in TSC infants (N=5).

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is caused by genetic mutation in TSC1 or TSC2, resulting in dysregulation of the mechanistic target of rapamycin (mTOR) signaling pathway. Age at time of seizure onset in TSC infants has been linked to long-term neurodevelopmental outcome in this high-risk population. TAVT-18 is a novel formulation of sirolimus, an mTOR inhibitor. This study evaluates TAVT-18 as a targeted, disease-modifying drug therapy for preventing or delaying seizure onset in TSC using a rational, mechanism-based therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* 0-6 months of age at the time of enrollment (randomization and treatment initiation must occur before 7 months of age and infants born prematurely must have a corrected age of at least 39 weeks, calculated by subtracting the number of weeks born before 40 weeks gestation from the actual chronological age, in weeks)
* Has a confirmed diagnosis of TSC based on established clinical or genetic criteria

Exclusion Criteria:

* Prior history of seizures (clinical or electrographic) at the time of enrollment or identified on baseline EEG
* Has been treated in the past or is currently being treated at the time of enrollment with conventional anticonvulsant medications (AEDs), systemic (oral) mTOR inhibitors (such as rapamycin, sirolimus, or everolimus), ketogenic-related special diet, or another anti-seizure therapeutic agent, device, or procedure
* Has taken any other investigational drug as part of another research study, within 30 days prior to the baseline screening visit
* Has a significant illness or active infection at the time of the baseline screening visit
* Has a history of significant prematurity, defined as gestational age <30 weeks at the time of delivery, or other significant medical complications at birth or during the neonatal period that other than TSC would convey additional risk of seizures or neurodevelopmental delay (i.e. HIE, severe neonatal infection, major surgery, prolonged ventilatory or other life-saving supportive care or procedures)
* Abnormal laboratory values at baseline (i.e., renal function, liver function, or bone marrow production) that are in the opinion of the investigator clinically significant and may jeopardize the safety of the study subject
* Prior, planned or anticipated neurosurgery within 3 months of the baseline visit
* Has a TSC-associated condition for which mTOR treatment is clinically indicated (i.e. SEGA or AML)
* Subjects who are, in the opinion of the investigator, unable to comply with the requirements of the study

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Krueger, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Masuda S, Lemaitre F, Barten MJ, Bergan S, Shipkova M, van Gelder T, Vinks S, Wieland E, Bornemann-Kolatzki K, Brunet M, de Winter B, Dieterlen MT, Elens L, Ito T, Johnson-Davis K, Kunicki PK, Lawson R, Lloberas N, Marquet P, Millan O, Mizuno T, Moes DJAR, Noceti O, Oellerich M, Pattanaik S, Pawinski T, Seger C, van Schaik R, Venkataramanan R, Walson P, Woillard JB, Langman LJ. Everolimus Personalized Therapy: Second Consensus Report by the International Association of Therapeutic Drug Monitoring and Clinical Toxicology. Ther Drug Monit. 2025 Feb 1;47(1):4-31. doi: 10.1097/FTD.0000000000001250. Epub 2024 Sep 25. PMID 39331837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participants were screened; all five were eligible for enrollment.
Groups:
- Stage 1 Open Label: Phase I/II, open-label PK and initial safety analysis. TAVT-18 administered orally twice daily to achieve precision dosing target of 10 ng/ml. Whole blood sirolimus levels are assessed at defined intervals on days 1, 7, and 14. After day 14, participants can elect to continue open-label treatment with TAVT-18 until 12 months of age. Final developmental outcomes are assessed at 24 months of age.
  TAVT-18 (sirolimus): The investigational drug product to be used in this study is TAVT-18, a proprietary formulation of sirolimus in clinical development, by Tavanta Therapeutics, Inc. It is provided in a powder formulation in pre-measured vials.
Period: Overall Study
Arm/Group | Stage 1 Open Label
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: months] | 2.0 [1.0 to 4.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety - Adverse Events
Description: Percentage of subjects reporting severe (CTCAE v5.0 grade >= 3) adverse event (AE) or serious adverse event (SAE)
Time Frame: 12 months of age
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
percentage of participants | 40

2. Primary Outcome: Efficacy - Time to Seizure Onset
Description: Time from treatment initiation to seizure onset
Time Frame: 12 months of age
Measure: Median (Full Range); unit: days
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 2
days | 102 [26 to 178]

3. Secondary Outcome: Treatment Discontinuance Due to Adverse Events
Description: Percentage of subjects that reduce or discontinue treatment due to an AE or SAE (any grade)
Time Frame: 12 months of age
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
percentage of participants | 20

4. Secondary Outcome: Treatment Disruption Due to Adverse Events
Description: Number of days treatment is withheld due to an AE or SAE (any grade).
Time Frame: 12 months of age
Measure: Median (Full Range); unit: days
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
days | 19.5 [0 to 54]

5. Secondary Outcome: Precision Dosing Accuracy
Description: Blood trough concentration of sirolimus (ng/ml)
Time Frame: 12 months of age
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 4
ng/mL | 6.6 [3.6 to 9.3]

6. Secondary Outcome: Age at Seizure Onset
Description: Patient age in months at time of seizure onset
Time Frame: 12 and 24 months of age
Measure: Median (Full Range); unit: months
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 3
months | 10.6 [2.9 to 19.7]

7. Secondary Outcome: Seizure Type
Description: Percentage of subjects reporting infantile spasms, focal seizures, or other seizure types
Time Frame: 12 and 24 months of age
Population: Five participants were enrolled in the study. Only three of the enrolled participants developed seizures during the course of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
percentage of participants
  12 months of Age -- Infantile Spasms | 40
  12 months of Age -- Focal Seizures | 20
  24 months of Age -- Infantile Spasms | 40
  24 months of Age -- Focal Seizures | 60

8. Secondary Outcome: Seizure Frequency
Description: Number of seizures in past 30 days
Time Frame: 12 and 24 months of age
Population: as for outcome 7
Measure: Number; unit: seizures
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
seizures
  12 months of Age | 0
  24 months of Age | 0

9. Secondary Outcome: TAND Severity Assessed by the TAND-L Checklist
Description: Overall severity rating on the TSC-associated Neuropsychiatric Disorders-Lifetime Version (TAND-L) Checklist. The TAND-L Checklist severity rating ranges from 0-10, with higher values indicating greater concern.
  Parent Rating: "Considering all of the issues reported today how much have these bothered, troubled, or distressed you/your child/family?"; Min = 0 Max = 10; higher values indicate greater concern.
  Clinician Rating: "Interviewer's judgement of impact/burden on the individual/child/family."; Min = 0 Max = 10; higher values indicate greater concern
Time Frame: 12 and 24 months of age
Population: All participants completed the assessment at 12 months of age. One participant was unable to complete the assessment at the 24 month timepoint.
Measure: Median (Full Range); unit: units on a scale (0 - 10)
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
units on a scale (0 - 10)
  12 months of Age -- Parent Rating | 2 [0 to 5]
  12 months of Age -- Clinician Rating | 2 [0 to 5]
  24 months of Age -- Parent Rating: number analyzed (Participants) | 4
  24 months of Age -- Parent Rating | 1 [0 to 2]
  24 months of Age -- Clinician Rating: number analyzed (Participants) | 4
  24 months of Age -- Clinician Rating | 3.5 [0 to 4]

10. Secondary Outcome: Adaptive Behavior Assessed by the the VABS
Description: Composite score on the Vineland Adaptive Behavior Scales (VABS). The VABS composite score is normed to 100 = average or 50% percentile in normal populations, with lower values indicative of greater concern.
  Adaptive Scale: Minimum = 20, Maximum = 140, Standard deviation is +/- 15
Time Frame: 12 and 24 months of age
Measure: Median (Full Range); unit: composite score
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
composite score
  12 months of Age -- Adaptive Behavior Composite Score | 91 [86 to 102]
  24 months of age -- Adaptive Behavior Composite Score | 88 [68 to 128]

11. Secondary Outcome: Global Neurodevelopment Assessed by the Bayley Scales of Infant Development
Description: Composite score on the Bayley Scales of Infant Development. The Bayley Scales of Infant Development is normed to 100 = average or 50% percentile in normal populations, with lower values indicative of greater concern.
  Cognitive Domain: Minimum = 40, Maximum = 160, Standard Deviation is +/- 15 Language Domain: Minimum = 40, Maximum = 160, Standard Deviation is +/- 15 Motor Doman: Minimum = 40, Maximum = 160, Standard Deviation is +/- 15
Time Frame: 12 and 24 months of age
Population: 24 months of Age: Cognitive Domain only four of five participants completed this assessment as one participant became ill during visit. Language and Motor Domains only three of five participants completed these assessments as one became ill during visit and one participant became non-compliant during testing.
Measure: Median (Full Range); unit: composite score
Arm/Group | Stage 1 Open Label
Number analyzed (Participants) | 5
composite score
  12 months of Age -- Cognitive Domain | 90 [70 to 110]
  12 months of Age -- Language Domain | 89 [75 to 100]
  12 months of Age -- Motor Domain | 87 [72 to 112]
  24 months of Age -- Cognitive Domain: number analyzed (Participants) | 4
  24 months of Age -- Cognitive Domain | 95 [70 to 100]
  24 months of Age -- Language Domain: number analyzed (Participants) | 3
  24 months of Age -- Language Domain | 77 [70 to 92]
  24 months of Age -- Motor Domain: number analyzed (Participants) | 3
  24 months of Age -- Motor Domain | 74 [74 to 87]

ADVERSE EVENTS:
Time Frame: 12 months of Age
Arm/Group | Stage 1 Open Label
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Open Label (N=5)
Constipation (Gastrointestinal disorders) | 2 (4) — Total Reported: 4; Grade 1: 4; Relatedness: Unrelated 100%
Excessive Flatulence (Gastrointestinal disorders) | 2 (4) — Total Reported: 4; Grade 1: 1; Grade 2: 3; Relatedness: Unrelated 100%
Emesis (vomiting) (Gastrointestinal disorders) | 1 (5) — Total Reported: 5; Grade 1: 5; Relatedness: Unrelated 100%
Hematochezia (Bloody stool) (Gastrointestinal disorders) | 1 (1) — Total Reported: 1; Grade 2: 1; Relatedness: Possibly related 100%
Diarrhea (Gastrointestinal disorders) | 1 (1) — Total Reported: 1; Grade 2: 1; Relatedness: Possibly related 100%
Stomatitis (mouth sores/ulcers) (Gastrointestinal disorders) | 2 (5) — Total Reported: 5; Grade 1: 2; Grade 2: 3; Relatedness: Probable 60%, Definite 40%
Pyrexia (fever) (General disorders) | 2 (8) — Total Reported: 8; Grade 2: 8; Relatedness: Unrelated 100%
Fussiness (General disorders) | 1 (13) — Total Reported: 13; Grade 1: 1, Grade 2: 12; Relatedness: Unrelated 100%
Discomfort/Pain due to Teething (General disorders) | 1 (3) — Total Reported: 3; Grade 2: 3; Relatedness: Unrelated 100%
Fatigue (General disorders) | 1 (1) — Total Reported: 1; Grade 1: 1; Relatedness: Unrelated 100%
Rash (Allergic reaction) (Immune system disorders) | 1 (1) — Total Reported: 1; Grade 2: 1; Relatedness: Unrelated 100%
Rhinitis (Infections and infestations) | 3 (4) — Total Reported: 4; Grade 1: 4; Relatedness: Unrelated 50%, Possible 50%
Otitis Media (Infections and infestations) | 3 (3) — Total Reported: 3; Grade 2: 3; Relatedness: Possible 66.7%, Probable 33.3%
Rhinosinusitis (Sinus infection) (Infections and infestations) | 1 (1) — Total Reported: 1; Grade 2: 1; Relatedness: Probable 100%
Abscess w/Infection (Infections and infestations) | 1 (1) — Total Reported: 1; Grade 2: 1; Relatedness: Unlikely 100%
Croup w/Stridor (Infections and infestations) | 1 (1) — Total Reported: 1; Grade 2: 1; Relatedness: Possible 100%
Respiratory Syncytial Virus (RSV) (Infections and infestations) | 1 (1) — Total Reported: 1; Grade 2: 1; Relatedness: Possible 100%
Hand-Foot-Mouth Disease (Infections and infestations) | 1 (1) — Total Reported: 1; Grade 2; Relatedness: Possible 100%
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (4) — Total Reported: 4; Grade 1: 2, Grade 3: 2; Relatedness: Definite 100%
Hypercholesterolemia (Metabolism and nutrition disorders) | 3 (4) — Total Reported: 4; Grade 1: 4; Relatedness: Definite 100%
Insomnia (Psychiatric disorders) | 2 (2) — Total Reported: 2; Grade 1: 1, Grade 2: 1; Relatedness: Unrelated 100%
Tussis (cough) (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Total Reported: 3; Grade 1: 2, Grade 2: 1; Relatedness: Unrelated: 66.7%, Possible: 33.3%
Rhinorrhea (Congestion) (Respiratory, thoracic and mediastinal disorders) | 2 (8) — Total Reported: 8; Grade 1: 4, Grade 2: 4; Relatedness: Unrelated 50%, Possible 50%
Lip Lesion (Skin and subcutaneous tissue disorders) | 1 (4) — Total Reported: 4; Grade 2: 4; Relatedness: Possible 100%
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (5) — Total Reported: 5; Grade 1: 4, Grade 2: 1; Relatedness: Unrelated 80%, Possible 20%
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) — Total Reported: 2; Grade 1: 2; Relatedness: Unrelated 100%
Hypertension (Vascular disorders) | 1 (1) — Total Reported: 1; Grade 2: 1; Relatedness: Unrelated 100%

LIMITATIONS AND CAVEATS:
Primary endpoints and universal treatment by study design continued through 12 months. Between 12-24 months, ongoing treatment with sirolimus was optional. In this study, 4/5 participants elected to continue sirolimus treatment through the secondary 24 month timepoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT04595513/Prot_SAP_000.pdf